CLINICAL TRIAL: NCT02134483
Title: Parathyroid Allo-transplantation With a New Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erhan Aysan (Other)
Responsible Party: Sponsor-Investigator, Erhan Aysan, Bezmialem Vakif University, SB Istanbul Education and Research Hospital
Organization: SB Istanbul Education and Research Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1234567; 79797979 (Registry Identifier: Bezmialem Vakif University)
Record Dates: First submitted 2014-05-01; First posted 2014-05-09 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Parathyroid Allo-transplantation
Keywords: Parathyroid; Permanent hypocalcemia; Transplantation

ARMS (1):
- Parathyroid allo-transplantation (Experimental): patients who have permanent hypoparatyroidism
  Interventions: Biological: Parathyroid allo-transplantation

INTERVENTIONS:
Biological: Parathyroid allo-transplantation — parathyroid allotransplantation with a new tecnique without immunosuppression

SUMMARY:
Parathyroid allo-transplantation (PA-t) is a valuable alternative in the treatment of permanent hypoparathyroidism. However, it is a difficult process that requires a number of trained staff and advanced laboratory equipment which bring high costs. In this study, we have identified a new PA-t technique.

DETAILED DESCRIPTION:
Hypoparathyroidism is a clinical problem which is associated with hypocalcemia, hyperphosphatemia, low parathyroid hormone levels and often manifests itself as a complication of thyroid surgery . Direct injury, ischemia or unintended excision of parathyroid tissue are the most common mechanisms that cause temporary or permanent hypoparathyroidism. Temporary hypoparathyroidism (<6 months) develops at 10% of cases after thyroid surgery and nearly half of them develops permanent hypoparathyroidism (>6 months) (3-5). Due to the rapid increase in thyroid cancer cases in recent years, total thyroidectomy and neck dissection is performed more frequently than before that yields increase in frequency of permanent hypoparathyroidism.

As a current standard treatment, oral or intravenous calcium preparations and active vitamin-D3 are used in the treatment of hypocalcemia which was developed due to permanent hypoparathyroidism (PH). However, this approach is a symptomatic treatment, must continue a lifetime, the cost is high and is only intended to correct hypocalcemia. Besides, it has no beneficial effect on metabolic problems due to PH.

For these reasons, less costly and effective treatments have been searched over 30 years and parathyroid allo-transplantation (PA-t) was introduced as a treatment alternative. Nonetheless, it did not meet the expectations completely. The main problem in PA-t is the development of immune and inflammatory response against graft tissue which shortens its life and impairs the efficacy of the treatment. Various kinds of treatment methods such as immunosuppression, microencapsulation and cultivation were tried to overcome this problem. Despite these treatment options, convincing results have not yet been achieved . In literature, PA-t cases are often presented as case reports, only a few clinical series are available .

In this study, we aimed to present the results of our new PA-t technique that is performed on 10 patients who were diagnosed as permanent hypocalcemia following thyroid surgery and had no benefit from standard medical therapy

ELIGIBILITY:
Inclusion Criteria:

* patients who have permanent hypocalcemia
* Patients who accept to participate to study

Exclusion Criteria:

-Patients who don't accept to participate to study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2015-05-01 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
to mesure patient's blood calcium | up to three months

SECONDARY OUTCOMES:
to mesure patient's parathormon levels | up to three months

OTHER OUTCOMES:
to control patient's need for calcium containing drugs | up to three months

CONTACTS AND LOCATIONS:
Overall Officials: erhan aysan, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Istanbul, Turkey (Türkiye)

REFERENCES:
- Available data/document: Article — https://www.ncbi.nlm.nih.gov/pubmed/26375142